CLINICAL TRIAL: NCT02849665
Title: Immediate Effect of Kangaroo Position in Electromyographic Activity and Microcirculation of Newborn Preterm: A Randomized Clinical Trial.
Brief Title: Immediate Effect of Kangaroo Position in Electromyographic Activity and Microcirculation of Newborn Preterm
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Professor Fernando Figueira Integral Medicine Institute (Other)
Responsible Party: Principal Investigator, Kaísa Trovão Diniz, It is PhD student in Mother and Child Health for Instituto de Medicina Integral Prof. Fernando Figueira (IMIP- Brazil ), where he earned a master's degree in the same area in 2012. Is currently Physiotherapist at IMIP., Professor Fernando Figueira Integral Medicine Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 458163/2014-7
Record Dates: First submitted 2016-07-26; First posted 2016-07-29 (Estimated); Last update posted 2017-08-16 (Actual); Status verified 2017-08

CONDITIONS: Child Development
Keywords: Kangaroo-Mother Care Method; child development

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Kangaroo Position (Experimental): The newborn remains in a vertical position, with limbs flexed, dressed in light clothes, maintaining skin-to-skin contact and the face on the adult's thorax.
  Interventions: Other: Kangaroo Position
- Not Kangaroo Position (No Intervention): The newborns will be not placed in the position Kangaroo.

INTERVENTIONS:
Other: Kangaroo Position
  Arms: Kangaroo Position

SUMMARY:
Introdution: The Kangaroo Mother Care is a perinatal care model for preterm and low weight newborn. The Kangaroo Position is the main feature of this method. The infant should be lightly dressed, in prone position and upright against the torax of the parents. Researches provides evidence that the Kangaroo Position induces an increase in myoelectric activity of preterm newborn. However, it is unknown how long the newborn should remain in the kangaroo Position so that ocurr changes in electromyographic. An increase in electromyographic activity was observed after 24 hours or more of submission to the Position Kangaroo, however period lower of submission to the Position Kangaroo have not been evaluated yet. Also unknown are the physiological mechanisms that cause this muscle response. One hypothesis would be the increase in temperature caused by skin to skin contact which could improve circulation in small vessels with direct influence on the infusion and nutrition of muscle tissue. Objective: Evaluate the immediate effect of Kangaroo position in the electromyographic activity and microcirculation of preterm newborn. Method: It will be a randomized and controlled trial from August 2016 to February 2017 with newborn preterm admitted at the Kangaroo Unit, IMIP. Newborns eligible according to the inclusion and exclusion criteria will be randomized into two groups: Kangaroo Group (experimental group) and Not Kangaroo Group (control group). The data of the electromyographic activity and the microcirculatory parameters will be assessed and recorded in three stages: before the Kangaroo position, one and three hours after of continuous submission in the Kangaroo Position (for the group of cases) and before the Kangaroo position, one and four after the three assessments (for the control group). In the control group, the preterm newborns will be not submitted to Kangaroo position until the completion of the last and third evaluation. The acquisition of the electromyographic signal will be conducted through an equipment electromyography Miotool 400® brand (Miotec Equipamentos Biomédicos - Brasil). To assess microcirculation will be used for the white light spectroscopy method through the drive moorVMS-OXY®. The project was submitted and approved by Ethics Committee for Research on Human Beings of IMIP (52381915.5.0000.5201). This study is part of a anchor project approved by Conselho Nacional de Desenvolvimento Científico e Tecnológico- CNPq (process 458163/2014-7).

ELIGIBILITY:
Inclusion Criteria:

* a gestational age of 27-34 weeks;
* corrected age of until 35 weeks at the time of the first examination;
* had not previously been in the kangaroo position;

Exclusion Criteria:

* Apgar lower than 7 in the 5th min;
* a history of grade III or IV intracranial haemorrhage (diagnosed by way of transfontanelar ultrasound and included in the medical records);
* seizures;
* congenital infections (cytomegalovirus, rubella, toxoplasmosis, syphilis and vertically transmitted HIV)
* malformations of the central nervous system (hydrocephaly and genetic syndromes), infections of the central nervous system (meningitis or encephalitis);
* congenital cardiopathy;
* traumas during delivery (injuries to the brachial plexus, dislocation of the hip and pelvis fractures) and gastro-oesophageal reflux disorder.

Ages: 27 Weeks to 35 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2016-10-01; Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Electromyographic activity | 15 minutes
  Measure of the changes in electric potential of muscle.
Tissue oxygen saturation - SO2 | 5 minutes
Relative oxygenated haemoglobin concentration - oxyHb | 5 minutes
Relative deoxygenated haemoglobin concentration - deoxyHb | 5 minutes
Relative total haemoglobin concentration -totalHb | 5 minutes
Temperature | 5 minutes
  Tissue temperature
Blood flow | 5 minutes
  A quantity proportional to the product of the average speed of the blood cells and their number concentration.

CONTACTS AND LOCATIONS:
Overall Officials: José E. Cabral Filho, PhD, Study Director — Instituto de Medicina Integral Prof. Fernando Figueira - IMIP; Rafael M. Miranda, PhD student, Study Chair — Instituto de Medicina Integral Prof. Fernando Figueira - IMIP; João G. Bezerra alves, PhD, Study Chair — Instituto de Medicina Integral Prof. Fernando Figueira - IMIP; Geraldine F. Clough, PhD, Study Chair — University of Southampton - Academic Unit of Human Development and Health; Kaísa T. Diniz, PhD student, Principal Investigator — Instituto de Medicina Integral Prof. Fernando Figueira - IMIP
Locations (1):
- Unidade Canguru, Recife, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Diniz KT, Cabral Filho JE, Miranda RM, Lima GMS, Figueredo NPDS, Araujo KFN. Short-time effect of the kangaroo position on electromyographic activity of premature infants: a randomized clinical trial. J Pediatr (Rio J). 2020 Nov-Dec;96(6):741-747. doi: 10.1016/j.jped.2019.10.003. Epub 2019 Oct 14. PMID 31622569